CLINICAL TRIAL: NCT03944278
Title: Pilot Evaluation of Thulium Laser Alone or in Combination With Broad Band Light for Treatment of Dermatologic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-18-TB01
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Dermatology/Skin - Other

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Thulium Device (Experimental): 1927 Laser Treatment
  Interventions: Device: Thulium Laser

INTERVENTIONS:
Device: Thulium Laser — Thulium laser for skin resurfacing procedures

SUMMARY:
Evaluate the Thulium laser device for skin resurfacing procedures, or as a treatment for pigmented lesions (age or sun spots) or dyschromia; or cutaneous lesions such as, but not limited to, actinic keratosis, melasma, fine rhytides; or as a method of improving skin tone and skin texture

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, 18 years and older
2. Fitzpatrick Skin Type I-VI
3. Subject has visible signs of moderate sun-damages and/or aging facial skin with visible areas of fine rhytides, pigmentation, and erythema or telangiectasia.
4. Desires non-ablative photo-revitalization of the skin.
5. Subject must agree to not make any changes in their skin regimen for the duration of the study, including the follow-up period.
6. Subject must be able to read, understand and sign the Informed Consent Form.
7. Must be willing and able to adhere to the treatment and follow-up schedule and post- treatment care instructions.
8. Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period.
9. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
10. Agree to not undergo any other procedure(s) in the treatment area during the study, such as laser- or light-based treatment, non-light based device treatment such as radiofrequency or ultrasound, injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler, chemical peel, or surgical procedure

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 3 months of study participation, such as laser or light-based procedures or surgery.
3. Prior injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler in the target area within 1 week of study participation.
4. History of malignant tumors in the target area.
5. Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
6. Pregnant and/or breastfeeding.
7. Having an infection, dermatitis or a rash in the treatment area.
8. Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
9. Suffering from coagulation disorders or taking prescription anticoagulation medications.
10. History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
11. History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
12. History of vitiligo, eczema, or psoriasis.
13. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
14. History of seizure disorders due to light.
15. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
16. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
17. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
18. History of pigmentary disorders, particularly tendency for hyper- or hypo- pigmentation.
19. Systemic use of retinoid, such as isotretinoin, or corticosteroid, as applicable, within 6 months of study participation.
20. Topical use of retinoid, such as isotretinoin, corticosteroid or hydroquinone on the target area within 1 month of participation.
21. Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
22. Excessively tanned in areas to be treated, or unable/unlikely to refrain from tanning during the study (for example, subject's occupation requires regular sun exposure).
23. Current smoker or history of smoking within 6 months of study participation.
24. Has infectious disease
25. Has been on long-standing systemic steroids (e.g. Prednisone, Dexamethasone)
26. Has medical condition that may affect wound healing
27. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Photography | 6 weeks post final treatment
  Change in photography when compared to baseline using Physicians global assessement scale

SECONDARY OUTCOMES:
Pain scores | Immediately after each treatment received
  Pain during treatment scored using Numeric pain scale 0-10, where 0 is least pain and 10 being maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Jay Patel, Study Director — Sciton
Locations (1):
- Refined Dermatology, Los Gatos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided